CLINICAL TRIAL: NCT04879680
Title: Indocyanine Green Fluorescence-guided Sentinel Node Biopsy in Breast Cancer Within a North African Population: a Retrospective Study
Status: Completed | Type: Observational
Sponsor: Faculty of Medicine, Sousse (Other)
Responsible Party: Principal Investigator, Samir Hidar, Prof. M.D, Faculty of Medicine, Sousse
Other Study IDs: CEFMS 82/2021
Record Dates: First submitted 2021-05-05; First posted 2021-05-10 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Breast Cancer; Sentinel Lymph Node
Keywords: breast cancer; sentinel node
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: sentinel node detection — Under general anesthesia 5 ml at 2.5mg/ml of Infracyanine ® (Laboratoire SERB; France) were injected circumferentially around the areola. Two ml of patent blue-V dye (Laboratoire Guerbet, Aulney-Sous-Bois, France) were injected in combination in the cohort of patients undergoing the procedure after primary chemotherapy. This was followed by a breast massage to facilitate absorption into the lymph vessels, then the surgical lights were turned off and image were obtained under near-infrared light using a first generation Near Infra Red (NIR) device [K]. Course of subcutaneous lymphatic drainage pathway fluorescence was followed up to where it disappeared to enter to deeper axilla and an incision was performed at that place. Lymphatic duct identification using the NIR camera allowed localization and removal of the sentinel lymph node(s).

SUMMARY:
Background Radio Isotopes and Blue dye alone or in combination are the most commonly used tracer agents in sentinel Node Biopsy for early breast cancer. Recent studies have found fluorescence method using Indo Cyanine Green as a promising technology with fewer disadvantages. This study represents the first within a North African setting.

Methods Retrospective analysis of our database that includes patients with clinically node-negative breast cancer scheduled for breast surgery and SN biopsy between 2016 and January 2021. Patients who underwent detection using fluorescence-ICG were included in this study.

DETAILED DESCRIPTION:
We performed a retrospective review our data base that includes breast cancer planned for sentinel node biopsy at the F. Hached University teaching hospital(Sousse, Tunisia). Data between April 2016 and January 2021 were reviewed. Only non-pregnant or lacting adult female patients without palpable clinical node and considered suitable for such procedure at multidisciplinary meeting were included. We excluded from our analysis the first ten cases considered as a learning curve Same operator (SH) carried out all the procedures.

Under general anesthesia 5 ml at 2.5mg/ml of Infracyanine ® were injected circumferentially around the areola. Two ml of patent blue-V dye (Laboratoire Guerbet, Aulney-Sous-Bois, France) were injected in combination in the cohort of patients undergoing the procedure after primary chemotherapy. This was followed by a breast massage to facilitate absorption into the lymph vessels, then the surgical lights were turned off and image were obtained under near-infrared light using a first generation Near Infra Red device . Course of subcutaneous lymphatic drainage pathway fluorescence was followed up to where it disappeared to enter to deeper axilla and an incision was performed at that place. Lymphatic duct identification using the NIR camera allowed localization and removal of the sentinel lymph node(s). Further fluorescent imaging was performed to identify potential residual signal in the axilla and such signal-sites were removed. Following ICG assisted-dissection, blue-stained nodes were excised if any. All detected sentinel node were send for frozen section and processed for histological examination. After sentinel node biopsy, conservative surgery or mastectomy were performed according to indication and axillary dissection was performed according to international guidelines.

Statistical analysis Baseline patient's and tumor characteristics, Identification Rate of the sentinel node with Indocyanine green and with dye , when used, were recorded. Data were entered and analyzed in Excel. The continuous variables are presented as mean ± standard deviation and categorical variables are presented as count and percentages unless specified. Informed consents from each patient and IRB approval were obtained

ELIGIBILITY:
Inclusion Criteria:

* non-pregnant or lacting adult female patients with breast cancer without palpable clinical node and considered suitable for such procedure at multidisciplinary meeting were included

Exclusion Criteria:

* Non eligible patient for breast cancer sentinel node procedure

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 47 patients who underwent SN biopsy using the above-mentioned technique were included. Mean age at time of surgery was 50.1 years (range 24-78 years).
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2021-03 (Actual); Study Completion 2021-04 (Actual)

PRIMARY OUTCOMES:
identification rate | 5 years
  percentage of cas in whom sentinel node was identified with fluoresence method

CONTACTS AND LOCATIONS:
Overall Officials: Samir Hidar, Prof. M.D, Principal Investigator — F.Hached university teaching hospital

IPD SHARING:
Plan to Share IPD: No